CLINICAL TRIAL: NCT02218437
Title: Child With Severe Aplastic Anemia (SAA) Therapy: the Injection of Umbilical Cord Derived Mesenchymal Stem Cells.
Brief Title: Treatment Protocol of Child SAA With the Injection of Mesenchymal Stem Cells（Umbilical Cord Derived）
Acronym: MSC-SAA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Xiaofan Zhu, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-2014-SAA-1; H0806-MSC-2014 (Other Grant/Funding Number: NSFC)
Record Dates: First submitted 2014-08-06; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Complications of Organ Transplant Stem Cells Umbilical Cord
Keywords: Mesenchymal Stem Cells (MSC); Umbilical Cord; thymocyte globulin (ATG); Severe Aplastic Anemia (SAA)
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC+ATG (Experimental): The first agent MSC injection, began two weeks after ATG application; Each patient was injected three times, one time per week; Study on single dose tolerance and efficacy index; Each subjects received three dose groups of treatment.
  Interventions: Drug: MSC+ATG

INTERVENTIONS:
Drug: MSC+ATG — MSC+ATG:Starting dose was 0.5-1.0 × 106 cells /kg; And the maximum tolerated dose was 1 ×107 cells /kg after ATG application.
  Other Names: Mesenchymal Stem Cells (Umbilical Cord Derived)

SUMMARY:
Mesenchymal Stem Cells (MSC) is a non Hematopoietic Stem Cells (HSC) in adult bone marrow and takes part in the bone marrow microenvironment. The response rate of early treatment on Children's SAA application combined with anti-thymocyte globulin (ATG) (40-50 days after ATG treatment) is associated with long-term effect. The injection of Umbilical Cord Derived Mesenchymal Stem Cells combined with ATG improves the efficacy of children with SAA.

DETAILED DESCRIPTION:
1. Mesenchymal Stem Cells were prepared by in vitro separation, screening, and culture from healthy human umbilical cord tissue; The " injection of mesenchymal stem cells (umbilical) manufacturing and verification regulation " was also formulated.
2. The starting dose of Umbilical Cord Derived MSC was 0.5-1.0 * 106 cells /kg, based on the previous human studies; And the maximum tolerated dose was 1 * 107 cells /kg
3. The response and complete remission rate, relapse rate of the injection of Umbilical Cord Derived Mesenchymal Stem Cells (or combined with ATG ) for Child with SAA were determined.

ELIGIBILITY:
Inclusion Criteria:

* Non-Severe Aplastic Anemia (NSAA)atients

Exclusion Criteria:

* Severe Aplastic Anemia (SAA) patients

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
The response and complete remission rate with different doses of Umbilical Cord Derived MSC to treat child with SAA | 1 year
  Complete response (CR) was defined as achieving normal levels of hemoglobin adjusted for age, platelet count >100*109/L, and absolute neutrophil count (ANC) >1.5*1.0 9/L. Partial response (PR) was defined as injection independence, reticulocyte count>30*109/L, platelet count >20*109/L, and ANC>0.5*1.0 9/L above the baseline. Persistence of injection requirement or death was evidence of no response (NR).

SECONDARY OUTCOMES:
The relapse rate with different doses of MSC to treat child with SAA | 3-10 year
  The relapse was defined as injection dependence again; or progressed or paroxysmal nocturnal hemoglobinuria (PNH)/acute myeloid leukemia/myelodysplasia syndrome(MDS); or cyclosporin A (CsA) dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, China

REFERENCES:
- [Derived] Lan Y, Liu F, Chang L, Liu L, Zhang Y, Yi M, Cai Y, Feng J, Han Z, Han Z, Zhu X. Combination of umbilical cord mesenchymal stem cells and standard immunosuppressive regimen for pediatric patients with severe aplastic anemia. BMC Pediatr. 2021 Feb 27;21(1):102. doi: 10.1186/s12887-021-02562-x. PMID 33639900